CLINICAL TRIAL: NCT04899388
Title: Pericapsular Nerve Group (PENG) Block Versus Lumbar Erector Spinae Plane Block as Postoperative Analgesia in Hip Surgeries: A Randomized Controlled Trial
Brief Title: Pericapsular Nerve Group (PENG) Block Versus Lumbar Erector Spinae Plane Block
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Marwa Mohamed Medhat, lecture of anesthesia and surgical intensive care (Principal Investigator), Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6818
Record Dates: First submitted 2021-03-19; First posted 2021-05-24 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Pericapsular Nerve Group Block (PENG Block); Lumbar Erector Spinae Plane Block
Keywords: Lumbar Erector Spinae Plane Block, Pericapsular Nerve Group Block (PENG Block)
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: douple
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PENG (Active Comparator): the patients lied in the supine position. The probe was originally placed in a transverse plane above the anterior superior iliac spine in the ipsilateral surgical site and then counterclockwise rotated about 45 degrees to line up with the pubic ramus. The iliopubic eminence, iliopsoas muscle and tendon, femoral artery, and pectineus muscle were all visible in this view. By an in-plane technique, from lateral to medial, a 22-gauge, 80-mm needle was placed in the musculofascial plane between both the psoas tendon anteriorly and the pubic ramus posteriorly .The local anesthetic medication was delivered after negative aspiration while looking out for proper fluid distribution for a total volume of 20 mL of Bupivacaine 0.25%
  Interventions: Procedure: Pericapsular Nerve Block
- ESPB (Active Comparator): TThe patient was positioned at the lateral decubitus posture in the ipsilateral surgical site. The convex USG transducer was moved from the midline to the side of the operation and positioned 4-6 cm lateral to the L3 spinous process in a longitudinal parasagittal plane. The needle was advanced using the in-plane superior-to-inferior approach. The needle was advanced with the tip introduced up to the plane anterior to the "erector spinae muscle" and the posterior surface of the L3 transverse process. 0.5-1 ml of normal saline was administered for hydrodissection and to ensure proper placement .If there was any resistance during administering local anesthesia, the needle was modified by drawing it back a few millimeters. the prepared local anesthetic solution 20 ml bupivacaine 0.25 % was delivered through the point between both the transverse process and the erector spinae muscle
  Interventions: Procedure: Lumbar Erector Spinae Plane Block
- control (Placebo Comparator): patients received spinal anesthesia without any block
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Procedure: Pericapsular Nerve Block — regional anaesthia
  Other Names: PENG
  Arms: PENG
Procedure: Lumbar Erector Spinae Plane Block — regional anaesthia
  Other Names: LESB
  Arms: ESPB
Drug: Fentanyl — intavenous
  Arms: control

SUMMARY:
assess and compare the efficacy of pericapsular nerve group block wersus lumber erector spinae plane block in reducing postoperative pain within the first 24 hours after hip surgeries.

DETAILED DESCRIPTION:
after being informed about the study and potential risks. All patients giving written consent will be randomized by double blind manner into 3groups each one containing 23 patients ,PENG group (n =23 ): The patients will receive Pericapsular Nerve Group Block (PENG Block) before positioning for spinal anesthesia.

ESPS group E (n =23 ): The patients will receive Lumbar Erector Spinae Plane Block before positioning for spinal anesthesia.

Control group C(n =23 ): patients received spinal anesthesia without any block.

ELIGIBILITY:
Inclusion Criteria:

Aged 65 to 75 years old. American Society of anesthesiologists physical status II and III. Body mass index of 25 to 30 kg/m2.

Exclusion Criteria:

Altered mental status. History of trauma or multiple fractures Uncontrolled hypertension and or diabetes. Coagulopathy. Preexisting advanced kidney, liver, or heart disease. Allergies or contraindications to the study drugs. Chronic use of opioids or corticosteroids.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
the time to first postoperative rescue analgesia | 24 hours postoperative
  the time to ask for the first postoperative analgesia (morphine) when the patient is reporting NRS ≥ 3

SECONDARY OUTCOMES:
Block performance time (min) | immediately before surgery
  time from placement of ultrasound probe on the patient's skin to the end of local anesthetic injection
onset of sensory block | after the block
  the time between the end of the injection of local anesthetic (bupivacaine) and the loss of pin prick sensation using a sterile 25G needle in the operating field.
pain intensity | 30 minutes after the end of surgery ,3,6,12 hours postoperative.
  using an 11point numeric rating scale (NRS)(11) : 0: no pain,10=worst imaginable pain) 1-3Mild Pain (nagging, annoying, interfering little with activities of daily living (ADLs).
  4-6Moderate Pain (interferes significantly with activities of daily living(ADLs) 7-10Severe Pain (disabling; unable to perform ADLs) at rest and during movement (during45-degree passive flexion of the hip with the ipsilateral knee flexed)
The total dose of rescue analgesia | 24 hours postoperative
  The total dose of rescue analgesia
adverse effects | 24 hours postoperative
  nausea, vomiting ,hypotension ,bradycardia and hematoma
Patient satisfaction | 24 hours postoperative
  related to block performance, post-operative pain relief was evaluated by an 11- point satisfaction score (0=unsatisfied and 10 = most satisfied), and the score was divided as follows 0-3 (not satisfied), 4-6 (partly satisfied), and 7-10 (highly satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Howida A kamal, M.D, Study Director — zagazig U; Marwa m Medhat, M.D, Principal Investigator — zagazig U
Locations (1):
- Aculty of Medicine,Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No